CLINICAL TRIAL: NCT07244120
Title: Effects of Embodied Writing Versus Conventional Writing Practice for Handwriting in Preschool Children.
Brief Title: Embodied Writing Versus Conventional Writing Practice for Handwriting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/AYESHAASIF
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Child Development
Keywords: Embodied writing, Conventional writing, HPSQ, MHA.

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial will involve 148 preschooler children of age group 3 to 6 years old with handwriting difficulties from Cambridge Foundation School FSD and Behan Je Memorial school FSD, Pakistan. The participants will be divided into two groups: Group A will follow conventional writing practices with parental ergonomics guidance, while Group B will engage in embodied writing practices combined with ergonomic education for parents. Over 8 weeks, handwriting legibility, speed, and motor coordination will be assessed pre- and post-intervention using the Handwriting Proficiency Screening Questionnaire and the Minnesota Handwriting Assessment Scale. The study aims to evaluate each approach's effectiveness in addressing handwriting challenges, providing insights into embodied learning's potential impact on early childhood education. Data analysis will be conducted using SPSS version 23.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both groups about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Conventional writing
  Interventions: Other: Conventional writing
- Group B (Active Comparator): Embodied writing
  Interventions: Other: Embodied writing

INTERVENTIONS:
Other: Conventional writing — Participants will perform: Tracing Patterns worksheets 5 repetitions of each for 15 min 3 times a week on alternate days for 8 weeks.Pencil Hold Exercises for Fingers:
  * Letter formation practice
  * Connecting Dots
  * Drawing Lines 5 repetitions of each for 25 min 3 times a week on alternate days for 8 weeks. 2. Guidelines about Correct Posture while writing will be given to Parents and class teacher.
    3. Post intervention assessment by tool MHA will use.
  Arms: Group A
Other: Embodied writing — Participants will involve whole body to perform these exercises:
  * Air Writing
  * Body Letter Shapes
  * Sand or Salt Tray tracing
  * Ribbon or Scarf writing 5 repetitions of each for 25 min 3 times a week on alternate days for 8 weeks.
  Obstacle course:
  * Balance Beam Letter (Walk along a beam or line on the floor, pausing to "write" a letter in the air or on a chalkboard at each end).
  * Letter Hopscotch (Hop between large letters drawn on the ground, calling out each letter's name or tracing its shape with a finger or a foot as they land on it).
  * Jump and Trace spots (Jump onto letter mats and trace the letter with fingers, a hand, or foot).5 repetitions of each for 15 min 3 times a week on alternate days for 8 weeks 3. Guidelines about Correct Posture while writing will be given to Parents and class teacher.
    4. Post intervention assessment by tool MHA will use.
  Arms: Group B

SUMMARY:
This randomized clinical trial will involve 148 preschooler children of age group 3 to 6 years old with handwriting difficulties from Cambridge Foundation School FSD and Behan Je Memorial school FSD, Pakistan. The participants will be divided into two groups: Group A will follow conventional writing practices with parental ergonomics guidance, while Group B will engage in embodied writing practices combined with ergonomic education for parents. Over 8 weeks, handwriting legibility, speed, and motor coordination will be assessed pre- and post-intervention using the Handwriting Proficiency Screening Questionnaire and the Minnesota Handwriting Assessment Scale. The study aims to evaluate each approach's effectiveness in addressing handwriting challenges, providing insights into embodied learning's potential impact on early childhood education. Data analysis will be conducted using SPSS version 23.

DETAILED DESCRIPTION:
This study explores the potential of embodied writing techniques to improve handwriting abilities in preschoolers, comparing it to traditional writing practices. Handwriting is foundational for cognitive development and academic performance, yet preschoolers often face challenges with it, stemming from issues in fine motor skills and coordination. Traditional writing methods typically emphasize structured exercises focused on repetitive tracing to enhance motor accuracy, but recent studies suggest that embodied writing learning through physical movement could offer unique benefits. By engaging the whole body, embodied writing encourages motor and cognitive engagement, helping children internalize movements and potentially improving both handwriting skills and overall learning engagement.

This randomized clinical trial will involve 148 preschooler children of age group 3 to 6 years old with handwriting difficulties from Cambridge Foundation School FSD and Behan Je Memorial school FSD, Pakistan. The participants will be divided into two groups: Group A will follow conventional writing practices with parental ergonomics guidance, while Group B will engage in embodied writing practices combined with ergonomic education for parents. Over 8 weeks, handwriting legibility, speed, and motor coordination will be assessed pre- and post-intervention using the Handwriting Proficiency Screening Questionnaire and the Minnesota Handwriting Assessment Scale. The study aims to evaluate each approach's effectiveness in addressing handwriting challenges, providing insights into embodied learning's potential impact on early childhood education. Data analysis will be conducted using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Child has poor handwriting as assessed by the HPSQ (20)
* Child is of age between 3-6 years.
* The child attends a regular primary school.
* Both boys and girls will be included in the study.

Exclusion Criteria:

* Developmental delay
* Physical impairment of upper extremity
* Hearing deficit (21)
* Visual problem
* Any recent trauma to upper limb
* Gross motor impairment
* Neurological deficit
* Receiving any Physiotherapy before

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Hand Proficiency Screening Questionnaire | Pre and post evaluation 1st week to 8th week
  The HPSQ-C can be used for a variety of academic and therapeutic purposes, including identifying handwriting deficiencies in school-aged children.An evaluation instrument called a handwriting proficiency screening questionnaire is used to gauge a person's handwriting abilities in a number of areas, including legibility, speed, motor control, and general handwriting quality. Its goal is to pinpoint issues or problems that could affect clear textual communication. It usually consists of questions about writing posture, grip, endurance, alignment, spacing, and letter formation. Teachers, therapists, and researchers frequently use this kind of questionnaire to evaluate children's or adults' handwriting skills. It can also be used as a preliminary screening tool to ascertain whether more thorough testing or intervention is required.

SECONDARY OUTCOMES:
Minnesota Handwriting Assessment MHA | Pre and Post evaluation 1st week to 8th week
  The MHA assesses children's handwriting skills by concentrating on five distinct areas: legibility, form, alignment, size, and spacing. Teachers and occupational therapists can use this evaluation to compare a child's handwriting skills to age-appropriate standards. The Minnesota Handwriting Test was created to satisfy occupational therapists' desire for a norm-referenced, educationally relevant assessment that could both identify pupils who struggle with handwriting and track the efficacy of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Asif, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenblum S, Gafni-Lachter L. Handwriting Proficiency Screening Questionnaire for Children (HPSQ-C): Development, Reliability, and Validity. Am J Occup Ther. 2015 May-Jun;69(3):6903220030. doi: 10.5014/ajot.2015.014761. PMID 25871594
- [Background] Klein E, Montgomery I, Zwicker JG. Evidence for pre-printing interventions: A scoping review. Journal of Occupational Therapy, Schools, & Early Intervention. 2021;14(4):400-36.